CLINICAL TRIAL: NCT00454831
Title: A 16 Week With 12 Week Active Treatment Multi-Center, Placebo-Controlled, Randomized Study Evaluating the Efficacy of HEP-40 Chitosan in Managing Moderate Hypercholesterolemia
Brief Title: Efficacy and Safety of HEP-40 Chitosan for Mild to Moderately Elevated Cholesterol
Acronym: HEP-40
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DNP Canada (Industry)
Collaborators: JSS Medical Research Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 153-PTL-001
Record Dates: First submitted 2007-03-30; First posted 2007-04-02 (Estimated); Last update posted 2007-11-16 (Estimated); Status verified 2007-11

CONDITIONS: Hypercholesterolemia
Keywords: Hypercholesterolemia; LDL-cholesterol; chitosan; HEP-40
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- HEP 400mg TID (Active Comparator): HEP-40 400 mg three times a day
  Interventions: Device: HEP-40 chitosan
- HEP 800mg BID (Active Comparator): HEP-40 800 mg twice a day
  Interventions: Device: HEP-40 chitosan
- HEP 800mg TID (Active Comparator): HEP-40 800 mg three times a day
  Interventions: Device: HEP-40 chitosan
- HEP 2400mg QD (Active Comparator): HEP-40 2400 mg once a day
  Interventions: Device: HEP-40 chitosan
- Placebo (Placebo Comparator): Placebo, three times a day
  Interventions: Device: HEP-40 chitosan

INTERVENTIONS:
Device: HEP-40 chitosan — Enzymatically Hydrolyzed Polychitosamine-40 kDa
  Other Names: Libracol

SUMMARY:
Chitosan is a natural product that is produced commercially through the deacetylation of chitin, which is found in the exoskeleton of crustaceans. It has been suggested that chitosan has a lipid-lowering effect.

This study was designed to determine if HEP-40 chitosan (Enzymatic Polychitosamine Hydrolysate - 40kDa), a short-chained chitosan with a molecular weight of 40 kDa, is safe and effective in lowering LDL-cholesterol levels in patients with mild to moderately elevated cholesterol levels and who have not been previously treated with other lipid-lowering agents.

DETAILED DESCRIPTION:
Chitosan is a natural product that is produced commercially through the deacetylation of chitin, which is found in the exoskeleton of crustaceans. It has been suggested that chitosan has a lipid-lowering effect by binding to fatty acids and cholesterol in the gastrointestinal tract and restricting their absorption.

This study was designed to determine if HEP-40 chitosan (Enzymatic Polychitosamine Hydrolysate - 40kDa), a short-chained chitosan with a molecular weight of 40 kDa, is safe and effective in lowering LDL-cholesterol levels in patients who have not been previously treated with lipid-lowering agents and who have cholesterol levels that are mild to moderately above the levels recommended by the National Cholesterol Education Program Adult Treatment Panel III (NCEP ATP III) guidelines.

This is a multi-centre, randomized, double-blind, placebo-controlled study. Following a 4-week Pre-Randomization Phase where patients will be instructed to maintain a stable diet, patients will be randomized to one of the following study groups for a 12-week Active Treatment Phase:

* HEP-40 400 mg three times a day (400 mg TID)
* HEP-40 800 mg twice a day (800 mg BID)
* HEP-40 800 mg three times a day (800 mg TID)
* HEP-40 2400 mg once a day (2400 mg QD)
* Placebo, three times a day (placebo)

The primary objective is to evaluate the clinical benefit of administering HEP-40 chitosan at different doses and at different dosing regimens compared with placebo. Clinical benefit will be defined as the reduction in LDL-cholesterol after 4 weeks of active treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with borderline, mild or moderate hypercholesterolemia, defined as LDL-C levels between 2.0 mmol/L and 4.5 mmol/L;
* At low (≤10%) or moderate (11-19%) 10-year risk for cardiovascular disease according to the Framingham model;
* Treatment-naïve for any lipid-lowering medications including statins, other pharmaceuticals or nutraceuticals;
* Stable diet and willing to continue on the dietary regimen recommended by their physician (NCEP Step 1 Diet) for the duration of the study;
* Woman of child bearing potential must be practicing effective birth control for a period of at least one month prior to initiation of the study.

Exclusion Criteria:

* Any concomitant condition which in the opinion of the investigator would preclude the patient from successfully participating in the study;
* Pregnant or that are breast feeding;
* Participation in another clinical trial within 30 days from initiation of the study;
* Known cardiac disease including: congestive heart failure, cardiac arrhythmias, unstable angina, myocardial infarction within the last 6 months, or uncontrolled malignant hypertension;
* High risk of developing coronary artery disease;
* Any condition affecting a major organ system, such as liver or kidney disease or malignancy;
* Uncontrolled diabetes mellitus or newly diagnosed patients (within 3 months) or recent change in anti-diabetic pharmacotherapy within 3 months of screening;
* Evidence of active renal disease indicated by serum creatinine > 2.0 mg/dL;
* Known HIV or Hepatitis B or C positive;
* Concurrent use of corticosteroids;
* Allergy or intolerance to crustaceans and/or seafood products.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2006-02; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Percent change in serum LDL-C between the baseline and 4-week visit compared to placebo. | 4 weeks

SECONDARY OUTCOMES:
Percent change in serum LDL-C from baseline to 8- and 12-weeks of treatment compared to placebo | 12 weeks
Percent change in serum total cholesterol from baseline to 12 weeks of treatment compared to placebo | 12 weeks
Percent change in serum HDL-C from baseline to 12 weeks of treatment compared to placebo | 12 weeks
Percent change in serum triglycerides from baseline to 12 weeks of treatment compared to placebo | 12 weeks
Safety and tolerability over the 12-week active treatment period, as determined by treatment-emergent adverse events. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jacques HF Lenis, MD, Principal Investigator — Recherche Invascor Inc; John S Sampalis, PhD, Study Director — JSS Medical Research Inc.
Locations (1):
- JSS Medical Research Inc., Westmount, Quebec, Canada